CLINICAL TRIAL: NCT02532296
Title: Improving Hospital-to-Home Care Transitions for High-risk Younger Adult Patients at a Safety Net Hospital: Activating Partnerships Among Patients, Families and Medical Staff
Brief Title: Improving Hospital-to-Home Care Transitions for High-risk Younger Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHA-3222
Record Dates: First submitted 2015-07-17; First posted 2015-08-25 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Patient Discharge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Receive usual hospital discharge, care transition and post-discharge care.
  Interventions: Behavioral: Control
- Transition Coach Intervention (Experimental): In addition to usual care, the intervention group receives care from a trained Transition Coach to support patients for 30 days after discharge.
  Interventions: Behavioral: Transition Coach (TC)

INTERVENTIONS:
Behavioral: Transition Coach (TC) — TC reviews patient's medical record to understand current admission and the medical/psycho-social history. TC makes introductory hospital visit(s) with patient to establish rapport and to define post-discharge needs.
  Starting in-house and continuing after discharge, TC helps patient set transition goals to maximize healthcare outcomes. Post-discharge, TC offers a voluntary face-to-face visit with patient along with weekly outreach calls, which are designed to assist patient with goal setting and attainment, medical system navigation; medication management; medical follow-up; transportation; use of community resources; and self-care.
  Intervention lasts 30 days post-discharge; afterwards TC seeks to handoff to an outpatient care team member, to ensure continuity of care.
  Arms: Transition Coach Intervention
Behavioral: Control — Receives usual hospital-based care, discharge preparation, transitional care and outpatient care.
  Arms: Control

SUMMARY:
Improving hospital-to-home care transitions can produce improvements in patient safety and health care outcomes, while decreasing medical costs. Most transitions research has examined strategies for older patients. This project, however, focuses on younger, high-risk patients within a safety net system. The proposed intervention is based on research that patient activation, as measured by the Patient Activation Measure (PAM), is correlated with risk for hospital readmission. The intervention seeks to increase PAM scores by employing a Transition Coach to coach patients, prior to and for 30-days after discharge, to (1) improve self-management skills through goal setting and goal attainment; (2) to enhance patient capacity to engage in trusting relationships with the Primary Care Provider (PCP), other medical specialists, family members of friends, and the Transition Coach; and (3) to improve ability to navigate the medical system.

The investigators will conduct a randomized trial to determine; (a) if PAM scores can be increased in the 30-day after hospital discharge; (b) if increased PAM scores, in this setting, are correlated with changes in healthcare utilization patterns; and (c) if the intervention presents a viable strategy to change healthcare utilization patterns and reduce rehospitalizations.

DETAILED DESCRIPTION:
Patient Activation is defined as the "knowledge, skills, confidence, and inclination to assume responsibility for managing one's health and healthcare needs." The 10-item version of the Patient Activation Measure (PAM) has been demonstrated to be a valid tool for measuring patient activation in a range of patient populations. Evidence demonstrates that PAM scores are correlated with heath care outcomes and that targeted interventions can modify PAM scores and improve outcomes.

Highly activated patients, based on their PAM scores, are less likely to experience 30-day readmissions, while those with lower levels of activation have higher rates of rehospitalization. The investigators propose an intervention to support younger adult patients transitioning from hospital to home to assume increased self-care responsibility. While hospitalization tends to promote the passive receipt of care, the intervention supports patients to take on a more active role. A Transition Coach will assist patients to prepare for discharge to enhance their ability to self-manage medications, follow-up appointments, symptoms, community services, and personal goals. The investigators hypothesize that intensified pre-discharge involvement in improving self-management skills for younger high-risk patients can; (a) improve PAM scores, (b) improve post-discharge engagement with medical, psychiatric and community-based care; and (c) present a strategy for changing healthcare utilization patterns that maximize outpatient care and reducing inpatient care, including hospital readmissions.

Patient Selection:

Cambridge Health Alliance (CHA) is a public safety-net system serving an ethnically diverse, underserved patient population of whom 30% are non-English speaking and 87% are publically insured. Our target group is high risk hospitalized medical patients age 60 and younger, who are discharged to home and receive primary care within the CHA network. Patients are considered high risk if they have had a previous inpatient admission or multiple Emergency Department (ED) visits within the past year, which serves as a proxy for complicated medical or psychosocial issues. Patients will be selected from the Medicine or Surgical Services at Cambridge Hospital.

Study Protocol:

The study protocol is described below.

1. The investigators anticipate enrolling 100 intervention patients and 100 control patients over 9 months.
2. A research assistant (RA) administers the Patient Activation Measure to intervention patients and control patients, immediately after randomization.

2- The intervention occurs with selected patients. 3- RA administers a post-discharge PAM to all patients 31 days after discharge.

Statistical Analysis:

Data will be extracted from the Electronic Medical Record (EMR) on all study patients. Baseline data will include age, sex, insurance status, Charlson comorbidity score, mental health and substance abuse disorders, marital status, homelessness, and address changes, admissions and ED visits in the past year.

Modest sample sizes may limit our ability to observe statistically significant effects. The PAM score is calculated with a scale of 0 to 100 (highest activation), with scores typically converted to a four-category categorical scale. Based on previous work in safety net settings,18 the investigators expect about 45% of control patients to have a PAM score of Level 4 (highly activated). With 100 intervention and 100 control patients, assuming two-sided alpha=0.05, the investigators would have 89% power to detect a 20% increase in the percentage of highly activated patients in the intervention group, and 65% power to detect a 15% increase. A key outcome is having an outpatient visit within 7 days of discharge. Based on our current work, only 15% of control patients in this group complete a 7-day visit. The investigators would have 81% power to detect an increase of 15% in the visit rate in the intervention group, and 50% power to detect a 10% increase.

Study Hypothesis:

The investigators expect to observe positive gains in PAM scores following the intervention, increases in 7-day outpatient follow-up rates and reductions in 30-day readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or less
* PCP within CHA network
* Have had at least one previous hospitalization or two or more Emergency Department visit within CHA in the past year
* Hospitalized at Cambridge Hospital on Medicine or Surgery Service
* Discharged from Medicine or Surgery service to home

Exclusion Criteria:

* Age > 60;
* Non-CHA PCP
* Discharged to rehabilitation or transferred to an outside hospital or to Psychiatry service

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline - Patient Activation Measure (PAM) and Utilization | 7,14, 30, 60, 90 days post-discharge
  Comparison between pre-discharge PAM and 30-day post-discharge PAM. Hospital and ED visit and outpatient visits with PCP and Specialists at 7,14,30,60,90 days.

SECONDARY OUTCOMES:
Goal Setting and Achievement | Hospital visit and 30 days post-discharge
  Number of goals defined and number of goals achieved
Relationship with Transition Coach (TC) | Hospital visit and 30 days post-discharge
  Number of encounters with TC (Hospital visits, Face-to-face visits, telephone outreach) and was TC acknowledged to be helpful in post-discharge period.
Relationship with PCP | 30 days post-discharge
  Number of PCP visits and was PCP acknowledged to be helpful in post-discharge period.
Relationship with other medical providers | 30 days post-discharge
  Number of specialty (non-psych) visit. Number of Psychiatric visits.
Relationship with Home Support | 30 days post-discharge
  Were friends or family acknowledged to be helpful in post-discharge period?
Ability to navigate health care system | 30, 60,180 days post-discharge
  Number of no-shows

OTHER OUTCOMES:
Pre-intervention utilization | 1 year pre-hospitalization
  ED visits, hospital admissions, outpatient visits, outpatient no-shows

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Balaban, MD, Principal Investigator — Cambridge Health Alliance
Locations (1):
- Cambridge Hospital, Cambridge, Massachusetts, United States